CLINICAL TRIAL: NCT05266339
Title: Cross-education in Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109
Record Dates: First submitted 2022-02-28; First posted 2022-03-04 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-06

CONDITIONS: Rotator Cuff Tears; Pain, Shoulder; Surgery
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cross-education group (Experimental): Each subject in the cross-education group will receive a treatment protocol consisting of cross-education (training of the contralateral limb) and standard exercise program applied after arthroscopic rotator cuff repair.
  Interventions: Other: Cross-education training; Other: Standard exercise program
- Standard exercise group (Active Comparator): Each subject in the standard exercise group will receive a treatment protocol consisting of standard exercise program applied after arthroscopic rotator cuff repair.
  Interventions: Other: Standard exercise program

INTERVENTIONS:
Other: Cross-education training — The strengthening exercises for rotator cuff muscles will be performed in the contralateral side of the affected side.
  Arms: Cross-education group
Other: Standard exercise program — The standard exercise program, which prepared according to The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation following arthroscopic rotator cuff repair, will be applied.

SUMMARY:
This randomized-controlled trial aims to investigate the efficacy of cross-education on function, pain, and range of motion, muscle strength and quality of life in patients who underwent arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Fifty voluntary patients who underwent arthroscopic rotator cuff repair, aged between 35-64 years will be randomly divided into two groups: Cross-education group and standard rehabilitation group. Interventions will be applied for 16 sessions (twice a week for 8 weeks). The patients will be assessed at baseline, at the end of the 8-week intervention and 1-month follow-up. The pain on activity, at rest and at night will be assessed with Visual Analog Scale (VAS). Active range of motion will be assessed with a digital goniometer. Isometric muscle strength will be measured with a handheld dynamometer. The functional status will be evaluated by Constant-Murley Score (CMS) and American Shoulder and Elbow Surgeons (ASES) Score. Health-related quality of life will be assessed with Short Form-12 (SF-12). The Global Rating of Change will be used to evaluate patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Being aged between 35-65 years Having undergone arthroscopic rotator cuff repair surgery Having the ability to read and write Turkish

Exclusion Criteria:

Revision surgery or previous shoulder surgery Having undergone subscapularis tendon repair in addition to arthroscopic rotator cuff repair Having scoliosis surgery or a health problem that will cause limitation in spinal mobility Restriction of movement or absence of limb in the opposite upper extremity Having frozen shoulder Presence of glenohumeral instability Having been diagnosed with thoracic outlet syndrome Presence of upper extremity fracture or tumor Having been diagnosed with cervical radiculopathy Having been diagnosed with any malignant condition, systemic, neurological or rheumatological disease Having a skin disease or hearing-vision problem that will affect the evaluation process

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score | Baseline
  The functional level will be assessed by the Constant Murley Score, which is a 100-point scale consisting of 15 points for pain, 20 points for daily activities, 40 points for pain-free range of motion, and 25 points for strength. High scores are positively correlated with the increased functional level. While pain and activities of daily living are evaluated by the patient, range of motion and strength are evaluated by the clinician.

SECONDARY OUTCOMES:
Constant-Murley Score | At the end of 8-week intervention
  The functional level will be assessed by the Constant Murley Score, which is a 100-point scale consisting of 15 points for pain, 20 points for daily activities, 40 points for pain-free range of motion, and 25 points for strength. High scores are positively correlated with the increased functional level. While pain and activities of daily living are evaluated by the patient, range of motion and strength are evaluated by the clinician.
Constant-Murley Score | 1-month follow-up after intervention
  The functional level will be assessed by the Constant Murley Score, which is a 100-point scale consisting of 15 points for pain, 20 points for daily activities, 40 points for pain-free range of motion, and 25 points for strength. High scores are positively correlated with the increased functional level. While pain and activities of daily living are evaluated by the patient, range of motion and strength are evaluated by the clinician.
Visual Analogue Scale | Baseline
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Visual Analogue Scale | At the end of 8-week intervention
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Visual Analogue Scale | 1-month follow-up after intervention
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Active Range of Motion Assessment | Baseline
  The shoulder flexion, abduction, internal and external rotation range of motion will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer. The process will be repeated three times in each direction, with the average value recorded.
Active Range of Motion Assessment | At the end of the 8-week intervention
  The shoulder flexion, abduction, internal and external rotation range of motion will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer. The process will be repeated three times in each direction, with the average value recorded.
Active Range of Motion Assessment | 1-month follow-up after intervention
  The shoulder flexion, abduction, internal and external rotation range of motion will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer. The process will be repeated three times in each direction, with the average value recorded.
Muscle Strength | At the end of the 8-week intervention
  Isometric muscle strength will be measured with a handheld dynamometer for shoulder flexion, abduction, internal and external rotation. The process will be repeated three times in each direction, with the average value recorded.
Muscle Strength | 1-month follow-up after intervention
  Isometric muscle strength will be measured with a handheld dynamometer for shoulder flexion, abduction, internal and external rotation. The process will be repeated three times in each direction, with the average value recorded.
American Shoulder and Elbow Surgeons Shoulder Score | Baseline
  The functional level will be measured using the American Shoulder and Elbow Surgeons Shoulder Score (ASES), which is created by the Society of the American Shoulder and Elbow Surgeons to facilitate standardization of outcome measures and to promote multicenter trials in shoulder and elbow surgery. This score contains a physician-rated and patient-rated section. The total score - 100 maximum points - is weighted 50% for pain and 50% for function.
American Shoulder and Elbow Surgeons Shoulder Score | At the end of the 8-week intervention
  The functional level will be measured using the American Shoulder and Elbow Surgeons Shoulder Score (ASES), which is created by the Society of the American Shoulder and Elbow Surgeons to facilitate standardization of outcome measures and to promote multicenter trials in shoulder and elbow surgery. This score contains a physician-rated and patient-rated section. The total score - 100 maximum points - is weighted 50% for pain and 50% for function.
American Shoulder and Elbow Surgeons Shoulder Score | 1-month follow-up after intervention
  The functional level will be measured using the American Shoulder and Elbow Surgeons Shoulder Score (ASES), which is created by the Society of the American Shoulder and Elbow Surgeons to facilitate standardization of outcome measures and to promote multicenter trials in shoulder and elbow surgery. This score contains a physician-rated and patient-rated section. The total score - 100 maximum points - is weighted 50% for pain and 50% for function.
Short Form-12 | Baseline
  Health-related quality of life will be assessed using the SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
Short Form-12 | At the end of the 8-week intervention
  Health-related quality of life will be assessed using the SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
Short Form-12 | 1-month follow-up after intervention
  Health-related quality of life will be assessed using the SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
Global Rating of Change | At the end of the 8-week intervention
  Patient satisfaction regarding improvement in shoulder function will be assessed by the Global Rating of Change (GRC) scale. The patients will be asked to rate their condition after a 8-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)